CLINICAL TRIAL: NCT01893099
Title: Sorafenib and Radioembolization With Sir-Spheres® for the Treatment of Metastatic Ocular Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Prof Olivier Michielin, M.D., Ph.D., Senior physician, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-CePO-code 16295
Record Dates: First submitted 2013-07-02; First posted 2013-07-08 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Ocular Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sorafenib- Cohort 1 (Experimental): Sorafenib 400 mg BID will be started 14 days after the administration of SIRT with SIR-Sphere®.
  Interventions: Drug: Sorafenib; Device: Radioembolization with SIR-Spheres® (Yttrium Microspheres)
- Sorafenib- Cohort 2 (Experimental): Sorafenib 400 mg BID will be started 11 days after the administration of SIRT with SIR-Sphere®.
  Interventions: Drug: Sorafenib; Device: Radioembolization with SIR-Spheres® (Yttrium Microspheres)
- Sorafenib- Cohort 3 (Experimental): Sorafenib 400 mg BID will be started 3 days after the administration of radioembolization with SIR-Sphere®.
  Interventions: Drug: Sorafenib; Device: Radioembolization with SIR-Spheres® (Yttrium Microspheres)
- Sorafenib- Cohort 4 (Experimental): Sorafenib 400 mg BID will be started 7 days prior to the administration of radioembolization with SIR-Spheres® and be given continuously, without drug holidays.
  Interventions: Drug: Sorafenib; Device: Radioembolization with SIR-Spheres® (Yttrium Microspheres)

INTERVENTIONS:
Drug: Sorafenib — Sorafenib will be given at the dosage of 400 mg BID. Initiation of the drug will vary dependently of the cohort and will be continued until progressive disease or intolerance.
  Other Names: Nexavar®
Device: Radioembolization with SIR-Spheres® (Yttrium Microspheres)

SUMMARY:
The best way to combine a loco-regional procedure such as chemoembolisation or radioembolization combined with an anti-angiogenic drug is not clear. This phase I trial aims to establish, first, the tolerability of the combination of liver radioembolization with SirSpheres® and sorafenib in uveal melanoma patients with liver metastasis studying different schedules of administration of sorafenib after and before radioembolization. Secondly, we aim to evaluate angiogenic markers modifications during these different schedules, either in the serum or radiologicaly. Dose of Sorafenib will be 400 mg BID and the timing of introduction will differ for one cohort to the other, given after the radioembolization for initials cohorts and finally, before and concomitantly to radioembolization for the last cohort.

DETAILED DESCRIPTION:
Primary objective:

To evaluate the safety and tolerability of sorafenib in combination with SIR-Spheres® radioembolization in uveal melanoma patients metastatic to the liver.

Secondary objectives:

* Translational research on biomarkers (blood and liver biopsies) as well as on radiological exam by using microbubble contrast enhanced ultrasound. Angiogenic markers such as VEGF, IGF-2, TFG Angiopoietin-2 and IL-8 will be monitored. Correlations will be investigated between the angiogenic markers (blood & tumor tissue), angiogenic radiological exam and the response to the treatment.
* To evaluate the response, clinical benefit, PFS and survival of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic uveal melanoma with proven histology (stage IV)
* Presence of liver metastases
* Concomitant non life-threatening metastases outside the liver are allowed
* Palliative radiotherapy will be allowed outside the liver
* Previous chemotherapy or immunotherapy at least 4 weeks before study treatment is allowed
* Age ≥ 18 years
* ECOG Performance Status of 0 or 1
* Life expectancy of at least 12 weeks
* Subjects with at least one uni-dimensional (by RECIST) measurable lesion. Lesions must be measured by CT-scan or MRI
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to study treatment

  * Hemoglobin ≥ 9.0 g/dl
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelet count ≥ 100,000/ul
  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN)
  * ALT and AST ≤ 5 x ULN
  * Alkaline phosphatase < 4 x ULN
  * PT-INR/PTT < 1.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN
  * Signed and dated informed consent before the start of specific protocol procedures

Exclusion Criteria:

* History of cardiac disease: congestive heart failure >NYHA class 2; active coronary artery disease (myocardial infarction more than 6 months prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension.
* History of HIV infection or chronic hepatitis B or C.
* Active clinically serious infections (> grade 2 NCI-CTC version 4.0).
* Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks before treatment start and is clinically stable with respect to the tumor at the time of study treatment).
* Patients with seizure disorder requiring medication (such as steroids or anti-epileptics).
* History of organ allograft.
* Patients with evidence or history of bleeding diasthesis.
* Patients undergoing renal dialysis.
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumor (Ta, Tis and T1) or any cancer curatively treated > 3 years prior to study treatment.
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test 72h before all investigations related to the protocol. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and two weeks after the completion of trial (and men for at least 3 months after last administration of study medication).
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study.
* Patients unable to swallow oral medications.
* Pre-treatment with any antiangiogenic agents (Bevacizumab, Sunitinib, or other TKI inhibitors affecting the vessels)
* Radiotherapy on the liver
* Major surgery within 4 weeks of start of treatment
* Autologous bone marrow transplant or stem cell rescue within 4 months of study treatment.
* Use of biologic response modifiers, such as G-CSF, within 3 weeks of study treatment.
* Investigational drug therapy outside of this trial during or within 4 weeks of study treatment
* Prior exposure to the study drug
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-06; Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Toxicity | 30 days of treatment of sorafenib
  Toxicities will be assessed according to the NCI-CTCAE (version 4.0).

SECONDARY OUTCOMES:
Translational research on biomarkers | 2 years
  Measurement of angiogenic factors and evaluation of angiogenesis with dynamic micro-bubble contrast-enhanced US
Clinical benefit | 2 years
  Clinical benefit (CR, PR and NC) evaluated with 18F-FDG-PET CT scan and CT scan by using respectively PERCIST criteria and RECIST criteria
Progression-free survival (PFS) | 2 years
Overall survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Michielin, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Derived] Berthod G, Cisarovsky C, Petrova T, Decosterd LA, Choong E, Celestini D, Cuendet MA, Boughdad S, Prior JO, Meuwly JY, Figg WD, Michielin O, Leyvraz S. Sorafenib plus selective internal radiotherapy with 90Y resin microspheres for the treatment of uveal melanoma with liver metastasis: a phase I trial. Br J Cancer. 2026 Feb;134(4):589-597. doi: 10.1038/s41416-025-03279-9. Epub 2025 Dec 11. PMID 41381843